CLINICAL TRIAL: NCT05314712
Title: Developing, Implementing, and Evaluating a Mixed-methods Community-based Participatory Research Sleep Intervention in Families With K-3rd Grade Children Living on the Blackfeet Indian Reservation
Brief Title: Assessing Sleep in Blackfeet Families With K-3rd Grade Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon Grant, Assistant Research Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VG032922; K01HL146993 (NIH)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Pre and post test of intervention group; pilot test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Intervention (Other): Pre and post test of 9-week intervention
  Interventions: Behavioral: Sleep intervention

INTERVENTIONS:
Behavioral: Sleep intervention — Participants will receive a 9-week sleep intervention through text and Facebook that include traditional Blackfoot cultural components combined with scientifically validated strategies for sleep.

SUMMARY:
This project will investigate traditional sleep routines and the current sleep environment in American Indian children to develop a culturally appropriate and novel sleep intervention to increase total sleep time for families with K-3rd grade children. The outcomes of this study will provide a comprehensive understanding of a relatively unknown behavior (sleep) in American Indians, show results from a novel sleep intervention in a high risk and underserved population, and will also contribute to the research and training development of an American Indian investigator, all defined missions of NHLBI.

DETAILED DESCRIPTION:
Children sleep less now than ever before. Despite a growing body of literature in understanding child sleep patterns, sleep interventions are limited. To date, there are no sleep intervention studies that have been done in AI tribal communities. Elders and community members play a critical role in identifying culturally adaptive solutions to address problems in tribal communities. Because of the prevalence of historical trauma and mistrust of outsiders, I am uniquely positioned to do this work in my own tribal community. Preliminary data of sleep patterns showed that Blackfeet children age 2-5 and age 12-15 averaged 10.15 hours and 7.5 hours of weekday sleep. Despite this understanding, evidence-based solutions to increase TST in tribal communities are unknown. Thus, I propose to explore traditional sleep routines coupled with asking Blackfeet families about the current sleep environment in their home to develop a culturally specific sleep intervention with one child and one adult dyad. I hypothesize that the sleep intervention will increase TST (primary outcome) in the dyads. The intervention may also result in improved physical activity and diet, and decreased stress and screen time (secondary outcomes). Data will be measured at 0 and 9 weeks and then at 3 month follow-up. This hypothesis will be tested in the following specific aims:

Specific Aim 1: Develop a culturally appropriate sleep intervention for Blackfeet families with K-3rd grade children using surveys, focus groups, interviews, community input, and evidence-based strategies on sleep.

Specific Aim 2: Feasibility test of the 9-week sleep intervention with K-3rd grade Blackfeet families.

The work proposed in these aims is designed to develop a comprehensive understanding of traditional sleep strategies and the child sleep environment to develop and pilot-test a novel culturally appropriate sleep intervention in the Blackfeet community. Developing culturally specific interventions to increase TST will address two significant gaps in the literature; understanding sleep problems in AI children and pilot-testing culturally adaptive sleep intervention strategies that will inform future research for investigators doing similar work in AI communities and provide direction for an R01 proposal that is one of the outcomes of this work.

ELIGIBILITY:
Inclusion Criteria:

• Blackfeet families with K-3rd grade children

Exclusion Criteria:

• Blackfeet families living off the Blackfeet Indian Reservation in Montana

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done through social media in the Blackfeet community. A total of 30 families (1 parent and 1 child) were recruited and consented. This was done summer and fall 2023.
Pre-assignment Details: As mentioned above, a total of 30 families were consented in the study. However, six families did not complete baseline data collection and a total of 14 families dropped out of the study. We were able to retain 23 families (46 parent/child dyads) for the study with post-intervention data on all participants.
Groups:
- Adult Participants; Child Participants: Pre and post test of 7-week intervention
  Sleep intervention: Participants will receive a 7-week sleep intervention through text and Facebook that include traditional Blackfoot cultural components combined with scientifically validated strategies for sleep.
Period: Overall Study
Arm/Group | Adult Participants | Child Participants
Started | 30 (We recruited a total of 30 families (60 participants overall; 30 adults) but only 23 adult participants completed baseline data collection.) | 30 (We recruited a total of 30 families (60 participants overall; 30 children) but only 23 child participants completed baseline data collection.)
Completed (A total of 14 participants dropped out of study.) | 23 | 23
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: All continuous data is represented as mean and standard deviation. All categorical data is number and percent.
Groups:
- Sleep Intervention: Pre and post test of 7-week intervention
  Sleep intervention: Participants will receive a 7-week sleep intervention through text and Facebook that include traditional Blackfoot cultural components combined with scientifically validated strategies for sleep.
Arm/Group | Sleep Intervention
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Adult age Population: There were 23 adult participants analyzed at baseline for age.
  years
    number analyzed (Participants) | 23
    (all) | 40.6 (13.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — Child Age Population: There were 23 child participants analyzed at baseline for age.
  years
    number analyzed (Participants) | 23
    (all) | 6.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Adult Participants Population: There were 23 adults analyzed at baseline for gender.
  Participants
    number analyzed (Participants) | 23
    Female | 21
    Male | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Child Participants Population: There were 23 children at baseline analyzed for gender.
  Participants
    number analyzed (Participants) | 23
    Female | 12
    Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Adult Participants Population: There were 23 adults analyzed at baseline for Race/Ethnicity
  Participants
    Blackfeet: number analyzed (Participants) | 23
    Blackfeet | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Child Participants Population: There were 23 children analyzed at baseline for Race/Ethnicity
  Participants
    Blackfeet: number analyzed (Participants) | 23
    Blackfeet | 23
Region of Enrollment [Number; unit: participants]
  United States | 46
Adult Height [Mean (Standard Deviation); unit: inches] — Height in inches Population: There were 23 adults measured at baseline for height
  inches
    number analyzed (Participants) | 23
    (all) | 66 (2.8)
Child Height [Mean (Standard Deviation); unit: inches] — Height in inches Population: There were 23 children at baseline measured for height.
  inches
    number analyzed (Participants) | 23
    (all) | 48.6 (9.9)
Adult Weight [Mean (Standard Deviation); unit: pounds] — Weight in pounds Population: There were 23 adults at baseline measured for weight
  pounds
    number analyzed (Participants) | 23
    (all) | 233.7 (51.1)
Child Weight [Mean (Standard Deviation); unit: pounds] — Weight in pounds Population: There were 23 children measured at baseline for weight
  pounds
    number analyzed (Participants) | 23
    (all) | 75.3 (41.4)
Adult Body Mass Index [Mean (Standard Deviation); unit: weight (kg)/height (m2)] — weight (kg)/height (m2) Population: There were 23 adults measured at baseline for BMI
  weight (kg)/height (m2)
    number analyzed (Participants) | 23
    (all) | 38.6 (8.2)
Child Body Mass Index [Mean (Standard Deviation); unit: weight (kg)/height (m2)] — weight (kg)/height (m2) Population: There were 23 children at baseline measured for BMI
  weight (kg)/height (m2)
    number analyzed (Participants) | 23
    (all) | 22.4 (5.7)
Adult Education [Count of Participants; unit: Participants] — Adults Education by high school, some college, and college degree Population: There were 23 adults at baseline measured for Education. This is not applicable to children.
  Participants
    number analyzed (Participants) | 23
    High School Diploma/GED | 6
    Some College/Associates Degree | 8
    College Degree | 9
Adult Income [Count of Participants; unit: Participants] — Adult income by catgeory Population: There were 23 adults measured at baseline for income. This is not applicable to children.
  Participants
    number analyzed (Participants) | 23
    $0-$20,000 | 4
    $21,000-$40,000 | 7
    $41,000-$60,000 | 6
    $61,000 or more | 6
Child Grade [Count of Participants; unit: Participants] — Number of children per grade Kindergarten through higher Population: There were 23 children at baseline measured for grade. This is not applicable to adults.
  Participants
    number analyzed (Participants) | 23
    Kindergarten | 7
    1st grade | 4
    Other | 12

OUTCOME MEASURES:

1. Primary Outcome: Sleep Trouble
Description: Sleep Trouble assessed by Pittsburgh Sleep Quality Index. Five questions on sleep trouble were asked on a likert scale that was treated as continuous and included four options: 0 = "Not during the past month"; 1 = "Less than a once a week"; 2 = "Once or twice a week"; 3 = "Three or more times a week." Each step in the scale represents an equal change on a continuous scale, e.g., going from a response of 1 to 2 is considered the same as going from 3 to 4. 0 is considered better and 3 is considered worse. The mean of the five responses were used as a total score for sleep trouble for each participant.
Time Frame: 7 weeks
Population: Adults sleep according to PSQI
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sleep Intervention
Number analyzed (Participants) | 23
Scores on a scale | 1.32 (0.53)
Statistical Analysis 1: Comparison: Sleep Intervention; Since all participants in this pilot study received in the intervention and data was collected pre and post intervention, there was no hypothesis test. Under the assumption that the likert scale data was treated as continuous, the data was analyzed using a linear mixed model. Variables in final model were included after variable selection (details below); Test type: Other — Linear Mixed Model (repeated measures model) of sleep trouble; There was no hypothesis test. All participants received the 7-week intervention - there was no comparison group. A variable selection approach (AIC) was used for including the final variables in the model; Using an exhaustive search of all models (dredge) that could be formed from predictor variables partner sleep rating, perceived stress, DASS scale, 8-item diet scale, amount of screen time, amount of time between bed time and wake time, amount of time to fall asleep, hours of sleep, sleep rating score, indicator variable if the child played outside, bed time, and wake time, adult height in inches, adult BMI, adult's highest education attained, the number of children in the household, grade of the child, child height in inches, child BMI, age of the child, and gender of the child, requiring the the timing of the survey be in the model, and accounting for repeated measurements over time, using AIC as the selection criterion we looked for the model with the smallest AIC value. The final sleep trouble model included the covariates timing of survey, DASS scale, and indicator variable if child played outside
Statistical Analysis 2: Comparison: Sleep Intervention; Since all participants in this pilot study received in the intervention and data was collected pre and post intervention, there was no hypothesis test. The data was analyzed using a mixed effects linear regression model. Variables in final model were included after variable selection (details below); Test type: Other — Mixed effects linear regression model of hours slept; [p-value comment as in outcome 1, analysis 1]; Using an exhaustive search of all models (dredge) that could be formed from predictor variables partner sleep rating, perceived stress, DASS scale, 8-item diet scale, amount of screen time, amount of time between bed time and wake time, amount of time to fall asleep, hours of sleep, sleep rating score, indicator variable if the child played outside, bed time, and wake time, adult height in inches, adult BMI, adult's highest education attained, the number of children in the household, grade of the child, child height in inches, child BMI, age of the child, and gender of the child, requiring the the timing of the survey be in the model, and accounting for repeated measurements over time, using AIC as the selection criterion we looked for the model with the smallest AIC value. The final model for hours slept included the covariates number of children in the household, indicator variable if child played outside, and baseline hours slept

ADVERSE EVENTS:
Time Frame: 7 weeks.
Description: The definition does not differ.
Arm/Group | Adult Participants | Child Participants
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT05314712/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT05314712/SAP_001.pdf
  • Informed Consent Form (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT05314712/ICF_002.pdf